CLINICAL TRIAL: NCT06350877
Title: One-on-one and Group-based Physical Activity Intervention Compared to a Wait-list Control for Post-secondary Student Mental Health and Well-being: A 3-arm Parallel Randomized Controlled Trial
Brief Title: 1:1 and Group-based Exercise Intervention for Post-secondary Student Mental Health and Well-being
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Melissa deJonge, Student Principal Investigator, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PA RCT
Record Dates: First submitted 2024-03-25; First posted 2024-04-08 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-04

CONDITIONS: Physical Activity; Mental Health Issue
Keywords: One-on-one physical activity; Group physical activity; Alternative mental health support; Mental health promotion
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: A 3-arm parallel Randomized Controlled Trial (RCT) assessing the immediate (post-intervention) and short-term (1-month) impact of the experimental arms (1:1 physical activity delivery and group-based physical activity delivery) compared to a 10-week control arm (wait-list control) will be conducted. A parallel arm design will be implemented, whereby participants will be randomized to a study arm and each study arm will be allocated a different intervention. The protocol adheres to CONSORT guidelines and SPIRIT recommendations for reporting of clinical trial protocols.
Who Masked: Care Provider
Masking Description: Following completion of the baseline assessment (T1), students will be randomly assigned to an experimental arm or the control arm by a program coordinator for the study. To prevent care provider bias, the physical activity coaches will remain blind to the purpose of group allocation and hypotheses of the study. Research Randomizer (www.randomizer.org) will be used to allocate participants into three equal groups using a blocked design (with an allocation ratio of 1:1:1).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 1:1 Physical Activity Intervention Delivery (Experimental): The physical activity intervention will be delivered using 1:1 coaching.
  Interventions: Behavioral: Physical Activity Intervention
- Group Physical Activity Intervention Delivery (Experimental): The group physical activity intervention will receive the physical activity intervention delivered in small groups of 3-8 students led by a trained sport and recreation coach.
  Interventions: Behavioral: Physical Activity Intervention
- 10-Week Waitlist Control Group (No Intervention): Students who are assigned to the 10-week waitlist control condition will be assessed on primary and secondary outcomes at baseline (T1), at 6-weeks (T2) and at 1-month follow-up (T3). At completion of the 1-month follow-up assessment, students in the wait-list control condition will be offered participation in the physical activity intervention; however, their behaviour will not be monitored or evaluated. Participants will have a choice of engaging in 1:1 physical activity intervention delivery or group-based physical activity intervention delivery.

INTERVENTIONS:
Behavioral: Physical Activity Intervention — The physical activity intervention will be a 6-week supervised program. Participation will involve engaging in a weekly 1-h session provided in-person at the campus athletics and recreation centre. Each 1-h session will include: (1) 30 min of behaviour change coaching; and (2) 30 min of supervised and structured physical activity training. The intervention materials will include a behaviour change workbook for facilitating the 30 min of behaviour change coaching. Each week participants will complete the behaviour change workbook in session with the program trainer, whereby the overarching goal is to introduce and reinforce engagement in behaviour change techniques and to facilitate the learning objectives and experiences for each weekly session.
  Arms: 1:1 Physical Activity Intervention Delivery; Group Physical Activity Intervention Delivery

SUMMARY:
Post-secondary students report alarming rates of feeling overwhelmed, hopeless, anxious, and depressed. To better support student mental health, there is a well-documented need to improve the range and quality of mental health services available to students. Focussing on formalized treatment approaches and strategies supporting well-being in the campus community more generally are needed. Physical activity is an alternative therapeutic approach that could be implemented as an evidence-based lifestyle intervention for supporting mental health and well-being on post-secondary campuses.

Despite the growing evidence supporting physical activity for student mental health, there are significant knowledge gaps in the literature. First, there is a paucity of research exploring the effects of different delivery styles (i.e., one-on-one (1:1) vs. group) on primary (i.e., mental health symptomology including anxiety symptoms, depression symptoms, psychological distress) and secondary (i.e., social support, social connectedness) outcomes. Secondly, the maintenance effects of a physical activity program on mental health or sustained physical activity behaviour change are largely unknown. Lastly, limited research has explored contextual implementation factors (e.g., intervention reach, adherence, and program satisfaction) that may influence the sustainability and scale-up of physical activity programs for student mental health. Examining contextual implementation factors is critical for optimizing physical activity intervention delivery and for facilitating wider dissemination of research findings into practice. The goal of this 3-arm parallel randomized controlled trial is to test the effectiveness of 1:1 physical activity intervention and group-based physical activity intervention compared to a wait-list control group in supporting post-secondary student mental health. The main questions include:

* Are there group differences between 1:1, group-based delivery, and waitlist control in the immediate (post-intervention) and follow-up (1-month) maintenance effects on the primary and secondary outcomes?
* Grounded in recommendations for process evaluation of complex interventions, what are contextual implementation factors that may be linked to variation in primary and secondary outcomes while offering insight for wider dissemination?

Trial participants will be randomly assigned to one of the following groups:

1. 1:1 physical activity training;
2. Group-based physical activity training consisting of small 5-8 person groups; or
3. Waitlist control. Students will participate in the physical activity intervention after the intervention and follow-up period (10 weeks); however, their participation will not be monitored or evaluated.

The physical activity training will involve a 6-week physical activity intervention consisting of weekly 1-hour sessions. Each session involves: (1) 30-minutes of behaviour change coaching (e.g., goal setting, action-planning, brainstorming strategies to overcome barriers to engaging in physical activity); and (2) 30-minutes of supervised and structured physical activity training. To address the aims of the study, participants will complete self-report questionnaires at baseline, post-intervention (following completion of the 6-week physical activity intervention), and 1-month following completion of the physical activity intervention. Questionnaires will assess demographic characteristics, primary outcomes (i.e., mental health symptomology including anxiety symptoms, depression symptoms, psychological distress), secondary outcomes (i.e., social support, social connectedness, physical activity behaviour) and contextual implementation factors (e.g., intervention reach, adherence, and program satisfaction) that may be linked to variation in primary and secondary outcomes while offering insight for wider dissemination. It is hypothesized that there will be no group differences between 1:1 delivery and group-based delivery on the primary outcomes. It is also hypothesized that group-based delivery, in comparison to 1:1 delivery will achieve greater improvements and more favourable maintenance effects in the secondary outcomes. Lastly, it is hypothesized that in comparison to the control group, 1:1 delivery and group-based delivery will be more effective in achieving change in the primary and secondary outcomes.

DETAILED DESCRIPTION:
Introduction

Post-secondary students report alarming rates of feeling overwhelmed, hopeless, anxious, and depressed. To better support student mental health, there is a well-documented need to improve the range and quality of mental health services available to students. Focussing on formalized treatment approaches and strategies supporting well-being in the campus community more generally are needed. Physical activity is an alternative therapeutic approach that could be implemented as an evidence-based lifestyle intervention for supporting mental health and well-being on post-secondary campuses.

Despite the growing evidence supporting physical activity for student mental health, there are significant knowledge gaps in the literature. First, research to date has predominantly been single-group designs with a lack of a control group and randomization. This contributes to limitations in the confidence and quality of the implications drawn from the synthesized studies. Indeed, within a post-secondary context, most studies are noted as poor quality and lack critical information regarding how they are designed, delivered, and made accessible to students. Second, there is a paucity of research exploring the effects of different delivery styles (i.e., one-on-one (1:1) vs. group) on primary (i.e., mental health symptomology reduction) and secondary (i.e., social support, social connectedness) outcomes. Importantly, group-based physical activity, in comparison to 1:1 delivered physical activity, may provide a less costly and less resource intensive intervention option, and may have unique benefits associated with exercising with others and peer-to-peer support (e.g., social support, a sense of belonging, expanded social networks). Third, the maintenance effects of a physical activity program on mental health or sustained physical activity behaviour change are largely unknown. As such, conclusions concerning achieving lasting change to mental health and sustained physical activity involvement are not possible. Lastly, limited research has explored contextual factors (e.g., intervention reach, adherence, and program satisfaction) that may influence the sustainability and scale-up of such programming opportunities. Examining contextual implementation factors is critical for optimizing physical activity intervention delivery and for facilitating wider dissemination of research findings into practice.

Objectives and Hypotheses

This randomized controlled trial study will assess the immediate (post-intervention, 6 weeks) and follow-up (4 weeks after post-intervention) maintenance effects of 1:1 supervised physical activity and group-based physical activity in comparison to a 10-week waitlist control group in reducing symptoms of poor mental health, supporting social well-being outcomes, and facilitating physical activity behaviour among post-secondary students experiencing poor mental health. The primary outcomes will be the immediate change in symptoms of poor mental health (anxiety symptoms, depression symptoms, psychological distress). The secondary outcomes will include follow-up change in symptoms of poor mental health (anxiety symptoms, depression symptoms, psychological distress) as well as the immediate and follow-up change in social well-being outcomes (social connectedness, social support), and physical activity behaviour. The aims of the study include: (1) examining group differences between 1:1 physical activity delivery, group-based physical activity delivery, and the 10-week waitlist control group on the primary and secondary outcomes; and (2) grounded in process evaluation recommendations, to explore contextual factors (e.g., intervention reach, adherence, and program satisfaction) that may be linked to variation in primary and secondary outcomes while offering insight for wider dissemination. It is hypothesized that there will be no group differences between 1:1 delivery and group-based delivery on the primary outcomes. It is also hypothesized that group-based delivery, in comparison to 1:1 delivery will achieve greater improvements and more favourable maintenance effects in the secondary outcomes. Lastly, it is hypothesized that in comparison to the control group, 1:1 delivery and group-based delivery will be more effective in achieving change in the primary and secondary outcomes.

Study Setting

The trial will be delivered in the post-secondary setting of a large metropolitan university. Importantly, post-secondary contexts offer natural advantages for large-scale implementation of physical activity programs for student mental health because they offer essential infrastructure (e.g., an integrated setting with access to sport and recreation facilities and mental health services) and practical support (e.g., experts in diverse fields) to develop, evaluate, and disseminate sustainable and scalable programs. Aligning with this perspective, the current study will employ a collaborative implementation approach, whereby the research team will work with on-campus sport and recreation professionals (i.e., for the provision of certified coaches with standard training in behavior change coaching and physical activity delivery) and mental health professionals in the post-secondary community (i.e., for program design, recruitment and implementation, and evaluation). In addition, purposeful efforts (e.g., through advocating for targeted referrals to the program and delivering targeted information sessions) will be made to promote the program among professionals (e.g., accessibility services, student-life services, health and wellness services) involved with providing mental health support or referrals to on-campus support services- an important approach for facilitating collaboration across disciplines and sectors in the campus community.

Participant Timeline

The university research ethics board (REB) has approved this study (protocol # 00045228). Students who meet eligibility and who have provided informed consent will be contacted to schedule an intake session with a program coordinator for the trial. Students who do not meet eligibility will be notified via email by the program coordinator and will be provided with a mental health resource sheet outlining alternative health and wellness programs and resources available to participate in. Intake sessions will be scheduled in-person in a private research space conveniently located in the campus athletics and recreation centre. During the intake session, participants will complete the baseline assessment (T1), and randomization will be conducted. Following completion of the intake session, participants in the experimental arms will complete the 6-week physical activity program (either 1:1 physical activity delivery or group-based physical activity delivery). In the experimental arms and control condition, study outcomes will be assessed at baseline (T1), 6-weeks post baseline (T2), and at 1-month follow-up (T3).

Sample Size

A 3 (group, individual, control) by 3 (T1, T2, T3) repeated measures design would require 25 participants per group assuming a moderate effect size of .30, a power level of .80, an alpha of .05, and expected correlations between timepoints of r = .50. To account for a loss to follow-up rate of 25%, the final targeted sample size is 93 post-secondary students. Participants will be randomly assigned to equal groups of approximately 31 students.

Recruitment

Purposive and snowball sampling procedures will be used to recruit post-secondary students who are physically inactive and experiencing poor mental health. Post-secondary students will be recruited and referred to the intervention through the team's research and professional networks (e.g., health and wellness and student support services; student life listservs; campus mental health listservs; the research team's social media platforms including Twitter and Instagram). Digital recruitment materials (including email scripts and poster advertisements) outlining the purpose of the intervention, intervention procedures, eligibility criteria, and a link to the screening questionnaire will be shared. The screening questionnaire will be administered through REDCap and allow participants to "sign up" up for the intervention through providing their email address and completing several screening questions to confirm eligibility. The program coordinator will contact eligible participants through their provided email address to confirm involvement in the study and to schedule an intake meeting.

Data Collection Methods

Statistical Methods

Preliminary analyses will include descriptive statistics (including mean scores for study variables, standard deviations, frequency counts for categorical variables and bivariate correlations) to examine the relationships between study variables and to describe participant characteristics. A 3 (group, individual, control) by 3 (T1, T2, T3) repeated measures ANOVA will be used to examine whether there are group differences between 1:1 physical activity delivery, group-based physical activity delivery, and the 10-week waitlist control group on the primary and secondary outcomes. Lastly, the implementation process evaluation outcomes will be assessed analyzing the responses to the closed-ended and open-ended questions. Closed-ended questions will be analyzed using descriptive statistics and open-ended questions will be analyzed using inductive thematic analysis.

Methods Monitoring

Harms

There are minimal risks or harms associated with participating in the research trial. Nonetheless, the current sample represents a population with relevant group vulnerability due to self-reported mental health concerns. There are also inherent risks associated with engaging in physical activity. First, it is possible that the self-report assessments may provoke negative emotions or may elicit uncomfortable thoughts and/or feelings. To mitigate emotional risks, participants will be informed of their right to not answer questions they feel uncomfortable answering, and all participants will be provided with a mental health resource sheet following completion of the intake meeting. Participants will also be informed of their right to withdraw from the trial without any penalty to their involvement in the 6-week physical activity intervention. Second, physical risks are rare but include cardiac events and musculoskeletal injuries. To reduce the risk of injury, the physical activity sessions will be delivered by certified sport and recreation coaches who have received standard training in behaviour change coaching and physical activity program delivery. Participants will also receive clearance for physical activity engagement using the PAR-Q+ and will be informed to refrain from engaging in any physical activity causing sharp pain, nausea, dizziness, or light-headedness. Bi-weekly meetings with the research team and sport and recreation coaches to mitigate any risks or concerns for participant vulnerability throughout the duration of the study will be held.

Ethics and Dissemination

Protocol Amendments

Protocol amendments, including but not limited to changes in the study objectives, the eligibility criteria, samples size, the outcomes, or statistical analyses will be submitted to appropriate REB review. Substantive changes will also be documented as amendments to the published study protocol and to the trial registry.

Confidentiality

All information collected for this trial will be kept strictly confidential. The information will be stored electronically in secure, password-protected folders only accessible to members of the research team. All data will be collected through a secure online data capture program (REDCap), where identifying information (i.e., email address, participant name) will be removed prior to data analysis. Data will be coded by participant ID and presented as aggregate-level data to maintain confidentiality and anonymity of the data.

ELIGIBILITY:
Inclusion Criteria:

* a post-secondary undergraduate or graduate student enrolled either part-time or full-time at a Canadian post-secondary institution
* fluent in English (e.g., proficiency in reading and verbal expression - written and oral)
* able to attend in-person physical activity sessions at the campus athletics and recreation centre
* moderately or insufficiently active ( < 23 units of weekly leisure activity) based on interpretation scores from the Godin Leisure-Time Physical Activity Questionnaire
* experiencing self-reported 'poor', 'fair' or 'good' mental health in the past month.

Exclusion Criteria:

* physically active (24 units or more of weekly leisure activity) based on interpretation scores from the Leisure-Time Physical Activity Questionnaire
* unsuccessful exercise clearance using the physical activity readiness questionnaire (PAR-Q)
* self-reported 'very good' or 'excellent' mental health

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Depression | T1 (0 days from baseline), T2 (42 days from baseline) T3 (72 days from baseline).
  To measure depression symptoms, the Participant Health Questionnaire will be used. The 9-item questionnaire measures the presence and severity of depressive symptoms over the past 2 weeks ranging from 0 (not at all) to 3 (nearly every day). The total summed score ranging from 0-27 will be used in main analyses
Anxiety | T1 (0 days from baseline), T2 (42 days from baseline) T3 (72 days from baseline).
  The Generalized Anxiety Disorder Questionnaire will be used to measure anxiety symptoms. The 7-item questionnaire assesses the frequency of symptoms associated with anxiety during the past two weeks ranging from 0 (not at all) to 3 (nearly every day). The total summed score ranging from 0-27 will be used in main analyses.
Psychological distress | T1 (0 days from baseline), T2 (42 days from baseline) T3 (72 days from baseline).
  Psychological distress will be measured using the 10-item Kessler Psychological Distress Scale. Students will be asked to indicate how often over the last 30 days they experienced symptoms of psychological distress ranging from 1 (none of the time) to 5 (all of the time). The total summed score (ranging from 10 - 50) will be used in analyses, with higher scores reflecting more psychological distress.
Well-being | T1 (0 days from baseline), T2 (42 days from baseline) T3 (72 days from baseline)
  The Mental Health Inventory-38 will be used to measure the 14-item psychological well-being subscale. Students will be asked to report how often during the past month they experienced symptoms of psychological well-being (e.g., How much of the time, during the past month, did you feel relaxed and free from tension; During the past month, how much of the time have you generally enjoyed the things you do?) on a six-point Likert scale. A total summed score will be used in main analyses, where higher scores represent more positive experiences of well-being.

SECONDARY OUTCOMES:
Social Connectedness | T1 (0 days from baseline), T2 (42 days from baseline) T3 (72 days from baseline).
  The 8-item Social Connectedness Scale will be used to measure social connectedness. The items portray a general emotional distance between the self and others and reflect behaviour, feelings, or both associated with a lack of connectedness on a 6-point Likert scale ranging from 1 (agree) to 6 (disagree). Scores will be reverse coded, thus higher scores will reflect a more reported sense of social connectedness with a potential range of 8-48.
Physical Activity Behaviour | T1 (0 days from baseline), T2 (42 days from baseline) T3 (72 days from baseline).
  Self-reported physical activity behaviour will be measured using the Godin Leisure-Time Exercise Questionnaire. Students will be asked to indicate how many times on average they engaged in mild (e.g., yoga, golf), moderate (e.g., fast walking, baseball), and vigorous (e.g., running, soccer) exercise for more than 15 minutes in a typical week. A common modification of assessing the average duration (in hours and minutes) per session of each intensity category of PA will be included (63-65). Students will also be asked to report the frequency and average duration of resistance exercise (e.g., free weight, bodyweight training). Total scores for mild, moderate, and vigorous activity and resistance exercise will be calculated by multiplying self-reported times per week by average duration of sessions for each type.
Social Support | T1 (0 days from baseline), T2 (42 days from baseline) T3 (72 days from baseline).
  To measure social support, the 5-item Social Provision Scale will be used. The scale consists of 5-items, on a 4-point Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree). A total summed score (ranging from 4 - 16) will be used in main analyses, where higher scores indicate more favorable perceptions of social support.
Intervention Reach | T2 (42 days from baseline)
  Intervention reach will be measured by descriptive data including recruitment and referral processes, the percentage of individuals who participate, the percent excluded, completion rates, and characteristics of participants compared with nonparticipants.
Therapeutic Alliance | T2 (42 days from baseline)
  Therapeutic alliance will be assessed using the 12-item Working Alliance Inventory. The Working Alliance Inventory has predominantly been studied and validated for use in psychotherapeutic contexts. Researchers, however, are increasingly supporting the importance of evaluating the coach-participant relationship for achieving favourable program outcomes. Participants will be asked to respond to each item on a 5-point Likert scale ranging from 1 (never) to 5 (always), wherein a higher score (ranging from 5 - 25) indicates a more positive therapeutic alliance.
Intervention Satisfaction | T2 (42 days from baseline)
  To assess intervention satisfaction a mix of closed-ended and open-ended questions will be used. The open-ended questions will assess general likes and dislikes towards the program and will be used to corroborate the closed-ended questions to provide an in-depth understanding of intervention satisfaction. Using closed-ended questions, students will be asked to self-report their physical activity session perceptions using 10-items on a 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree), with higher scores indicating more positive evaluations. Items will be treated as singular continuous variables, and descriptively analyzed.
Coach Perceptions | T2 (42 days from baseline)
  Participants will be asked to respond to 14-items on a 7-point Likert scale from 1 (Strongly disagree) to 7 (Strongly agree) assessing perceptions of the physical activity coach's ability to integrate core components of the program including providing a supportive environment, taking into account individual needs and preferences, and promoting engagement in enjoyable physical activity options. Higher scores ranging from 14 - 49 will indicate more favourable coach perceptions. Items will be treated as singular continuous variables, and descriptively analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Toronto, Mental Health and Physical Activity Research Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] American College Health Association. American College Health Association-National College Health Assessment II: Canadian Consortium Executive Summary Spring 2019. 2019. https://www.cacuss.ca/files/Research/NCHA-II%20SPRING%202019%20CANADIAN%20REFERENCE%20GROUP%20EXECUTIVE%20SUMMARY.pdf
- [Background] Andermo S, Hallgren M, Nguyen TT, Jonsson S, Petersen S, Friberg M, Romqvist A, Stubbs B, Elinder LS. School-related physical activity interventions and mental health among children: a systematic review and meta-analysis. Sports Med Open. 2020 Jun 16;6(1):25. doi: 10.1186/s40798-020-00254-x. PMID 32548792
- [Background] Ashdown-Franks G, deJonge M, Arbour-Nicitopoulos KP, Sabiston CM. Exploring the feasibility and acceptability of a physical activity programme for individuals with serious mental illness: A case study. Qualitative Research in Sport, Exercise, and health. 2022; 14(6): 933-955. doi:10.1080/2159676X.2021.2019098
- [Background] Barnett P, Saunders R, Buckman JEJ, Cardoso A, Cirkovic M, Leibowitz J, Main N, Naqvi SA, Singh S, Stott J, Varsani L, Wheatly J, Pilling S. Are students less likely to respond to routinely delivered psychological treatment? A retrospective cohort analysis. Compr Psychiatry. 2022 Nov;119:152348. doi: 10.1016/j.comppsych.2022.152348. Epub 2022 Sep 29. PMID 36191389
- [Background] Braun V, Clarke, V. Using thematic analysis in psychology. Qualitative research in psychology. 2006; 3(2): 77-101.
- [Background] Carter T, Guo B, Turner D, Morres I, Khalil E, Brighton E, Armstrong M, Callaghan P. Preferred intensity exercise for adolescents receiving treatment for depression: a pragmatic randomised controlled trial. BMC Psychiatry. 2015 Oct 14;15:247. doi: 10.1186/s12888-015-0638-z. PMID 26467764
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Background] Cornish PA, Berry G, Benton S, Barros-Gomes P, Johnson D, Ginsburg R, Whelan B, Fawcett E, Romano V. Meeting the mental health needs of today's college student: Reinventing services through Stepped Care 2.0. Psychol Serv. 2017 Nov;14(4):428-442. doi: 10.1037/ser0000158. PMID 29120201
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] deJonge ML, Omran J, Faulkner GE, Sabiston CM. University students' and clinicians' beliefs and attitudes towards physical activity for mental health. Mental Health and Physical Activity. 2020; 18. doi: 10.1016/j.mhpa.2019.100316
- [Background] deJonge ML., Jain S, Faulkner GE, Sabiston CM. On campus physical activity programming for post-secondary student mental health: Examining effectiveness and acceptability. Mental Health and Physical Activity. 2021; 20. doi: 10.1016/j.mhpa.2021.100391
- [Background] Gaglio B, Shoup JA, Glasgow RE. The RE-AIM framework: a systematic review of use over time. Am J Public Health. 2013 Jun;103(6):e38-46. doi: 10.2105/AJPH.2013.301299. Epub 2013 Apr 18. PMID 23597377
- [Background] Godin G. The Godin-Shephard Leisure-Time Physical Activity Questionnaire. The Health and Fitness Journal of Canada. 2011; 4(1): 18-22. doi: 10.4288/hfjc.v4i1.82
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Hunt J, Eisenberg D. Mental health problems and help-seeking behavior among college students. J Adolesc Health. 2010 Jan;46(1):3-10. doi: 10.1016/j.jadohealth.2009.08.008. Epub 2009 Oct 20. PMID 20123251
- [Background] Jeftic I, Furzer BJ, Dimmock JA, Wright K, Boyd C, Budden T, Rosenberg M, Kramer B, Buist B, Fitzpatrick I, Sabiston C, de Jonge M, Jackson B. Structured exercise programs for higher education students experiencing mental health challenges: background, significance, and implementation. Front Public Health. 2023 Apr 25;11:1104918. doi: 10.3389/fpubh.2023.1104918. eCollection 2023. PMID 37181716
- [Background] Jeftic I, Furzer B, Dimmock JA, Wright K, Budden T, Boyd C, Simpson A, Rosenberg M, Sabiston CM, deJonge M, Jackson B. The Stride program: Feasibility and pre-to-post program change of an exercise service for university students experiencing mental distress. Psychol Sport Exerc. 2023 Nov;69:102507. doi: 10.1016/j.psychsport.2023.102507. Epub 2023 Aug 16. PMID 37665942
- [Background] Jetten J, Haslam C, von Hippel C, Bentley SV, Cruwys T, Steffens NK, Haslam SA. "Let's get physical" - or social: The role of physical activity versus social group memberships in predicting depression and anxiety over time. J Affect Disord. 2022 Jun 1;306:55-61. doi: 10.1016/j.jad.2022.03.027. Epub 2022 Mar 14. PMID 35301039
- [Background] Kessler RC, Andrews G, Colpe LJ, Hiripi E, Mroczek DK, Normand SL, Walters EE, Zaslavsky AM. Short screening scales to monitor population prevalences and trends in non-specific psychological distress. Psychol Med. 2002 Aug;32(6):959-76. doi: 10.1017/s0033291702006074. PMID 12214795
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Litwiller F, White C, Hamilton-Hinch B, Gilbert R. The impacts of recreation programs on the mental health of postsecondary students in North America: An integrative review. Leisure Sciences. 2021; 44(1). doi: 10.1080/01490400.2018.1483851
- [Background] Lee RM, Robbins SB. Measuring belongingness: The Social Connectedness and the Social Assurance scales. Journal of Counseling Psychology. 1995; 42(2):232-241. doi: 10.1037/0022-0167.42.2.232
- [Background] Moore GF, Audrey S, Barker M, Bond L, Bonell C, Hardeman W, Moore L, O'Cathain A, Tinati T, Wight D, Baird J. Process evaluation of complex interventions: Medical Research Council guidance. BMJ. 2015 Mar 19;350:h1258. doi: 10.1136/bmj.h1258. PMID 25791983
- [Background] Muir IL., Munroe-Chandler KJ, Loughead TM, Sutherland CA, & Hawksley KG.The uworkitout uwin program: Improving university students' psychological distress through physical activity. International Journal of Kinesiology and Sports Science. 2020; 8(3). doi: 10.7575/AIAC.IJKSS.V.8N.3P.36
- [Background] Nesbitt AE, Collins KJ, Nalder E, Sabiston CM. Occupational Outcomes of a Physical Activity Intervention for Post-Secondary Student Mental Health. Can J Occup Ther. 2021 Sep;88(3):254-265. doi: 10.1177/00084174211021708. Epub 2021 Jun 16. PMID 34132119
- [Background] Okanagan Charter. Okanagan Charter: An International Charter for Health Promoting Universities & Colleges. 2015. https://wellbeing.ubc.ca/okanagan-charter
- [Background] Orpana HM, Lang JJ, Yurkowski K. Validation of a brief version of the Social Provisions Scale using Canadian national survey data. Health Promot Chronic Dis Prev Can. 2019 Dec;39(12):323-332. doi: 10.24095/hpcdp.39.12.02. PMID 31825785
- [Background] Pascoe M, Bailey AP, Craike M, Carter T, Patten R, Stepto N, Parker A. Physical activity and exercise in youth mental health promotion: a scoping review. BMJ Open Sport Exerc Med. 2020 Jan 23;6(1):e000677. doi: 10.1136/bmjsem-2019-000677. eCollection 2020. PMID 32095272
- [Background] Rebar AL, Stanton R, Geard D, Short C, Duncan MJ, Vandelanotte C. A meta-meta-analysis of the effect of physical activity on depression and anxiety in non-clinical adult populations. Health Psychol Rev. 2015;9(3):366-78. doi: 10.1080/17437199.2015.1022901. Epub 2015 Jul 3. PMID 25739893
- [Background] Sampson K, Priestley M, Dodd AL, Broglia E, Wykes T, Robotham D, Tyrrell K, Ortega Vega M, Byrom NC. Key questions: research priorities for student mental health. BJPsych Open. 2022 May 10;8(3):e90. doi: 10.1192/bjo.2022.61. PMID 35535504
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomized trials. Ann Intern Med. 2010 Jun 1;152(11):726-32. doi: 10.7326/0003-4819-152-11-201006010-00232. Epub 2010 Mar 24. PMID 20335313
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Stubbs B, Vancampfort D, Rosenbaum S, Ward PB, Richards J, Soundy A, Veronese N, Solmi M, Schuch FB. Dropout from exercise randomized controlled trials among people with depression: A meta-analysis and meta regression. J Affect Disord. 2016 Jan 15;190:457-466. doi: 10.1016/j.jad.2015.10.019. Epub 2015 Oct 29. PMID 26551405
- [Background] Stubbs B, Vancampfort D, Hallgren M, Firth J, Veronese N, Solmi M, Brand S, Cordes J, Malchow B, Gerber M, Schmitt A, Correll CU, De Hert M, Gaughran F, Schneider F, Kinnafick F, Falkai P, Moller HJ, Kahl KG. EPA guidance on physical activity as a treatment for severe mental illness: a meta-review of the evidence and Position Statement from the European Psychiatric Association (EPA), supported by the International Organization of Physical Therapists in Mental Health (IOPTMH). Eur Psychiatry. 2018 Oct;54:124-144. doi: 10.1016/j.eurpsy.2018.07.004. PMID 30257806
- [Background] Teychenne M, White RL, Richards J, Schuch FB, Rosenbaum S, Bennie JA. Do we need physical activity guidelines for mental health: What does the evidence tell us? Mental Health and Physical Activity. 202; 18: 100315. doi: 10.1016/j.mhpa.2019.100315
- [Background] Tracey TJ, Kokotovic AM. Factor structure of the Working Alliance Inventory. Psychological Assessment. 1989; 1(3): 207-210. doi: 10.1037/1040-3590.1.3.207
- [Background] Warburton DER, Jamnik VK, Bredin SSD, Gledhill N. The Physical Activity Readiness Questionnaire for Everyone (PAR-Q+) and Electronic Physical Activity Readiness Medical Examination (ePARmed-X+). Health and Fitness Journal of Canada. 2011; 4(2): 3-17.
- [Derived] deJonge ML, Yuen S, Simard L, Sabiston CM. One-on-one and group-based physical activity intervention compared to a waitlist control for post-secondary student mental health and social well-being: A 3-arm parallel randomized controlled trial protocol. PLoS One. 2025 Aug 29;20(8):e0330851. doi: 10.1371/journal.pone.0330851. eCollection 2025. PMID 40880346